CLINICAL TRIAL: NCT03492840
Title: An Open Label, Phase 2a Clinical Trial for the Evaluation of Safety and Efficacy of RZL-012 for the Treatment of Women With Lipedema Involving Substantial Fat Above the Knee or of Women and Men With Nodular Dercum's Disease
Brief Title: Treatment of Women With Lipedema Involving Substantial Fat Knee of Women and Men With Nodular Dercum's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RZL-012-FD-P2aUS-001.70; NCT04076891 (obsolete NCT alias)
Record Dates: First submitted 2018-02-19; First posted 2018-04-10 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2019-04

CONDITIONS: Lipedema; Dercum Disease
MeSH Terms: conditions — Lipedema; Adiposis Dolorosa | interventions — RZL-012

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Dercum's Disease (Active Comparator): Nodular size - diameter (cm) 2-2.9, 3-3.9, 4-8 Total dose of RZL-012(mg) 10 15 20 Dose per NOAEL 1/25th , 1/18.75th, 1/12.5th Number of injections: 2,3,4
  Interventions: Drug: RZL-012
- Cohort 2 - Lipedema (Active Comparator): Total dose of RZL-012 (mg) 60 , 80 Dose per NOAEL: 1/4.6888, 1/3.125 Number of injections: 12, 16
  Interventions: Drug: RZL-012

INTERVENTIONS:
Drug: RZL-012 — The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites

SUMMARY:
This is an open label, 2 cohort, clinical trial in women with lipedema with substantial fat above the knee and men with Dercum's disease. Each cohort will have 6 subjects who will receive RZL-012.

DETAILED DESCRIPTION:
This is an open label, 2 cohort, clinical trial in women with lipedema with substantial fat above the knee and men with Dercum's disease.

* The 1st cohort will be comprised of subjects with Dercum's disease.
* The 2nd cohort will be comprised of subjects with lipedema with substantial fat above the knee

Within each cohort dosing of the subjects will progress consecutively from one individual to the other with a minimum 7 days between subjects to asses safety. The study design will allow the physicians to monitor safety for at least 7 days prior to dosing the next subject. Cohort 2 will be conducted in a dose escalation manner and the decision to proceed to the next dose level will be made after reviewing all safety data collected by Day 14 within 2+/-1 day of the last dosed subject. The trial will proceed within a cohort provided that no more than one subject experience intolerable side effects in a cohort, and based on the decision made by the Principal Investigator (PI) and the medical monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal (at least 2 years) women no more than 65 years old, with lipedema involving substantial fat above the knee or nodular Dercum's disease in such women and in men 20 - 65 years with nodular Dercum's disease.
2. For Dercum's disease subjects - at least 2 nodules to be injected of at least 2cm diameter each, as determined by ultrasound
3. For lipedema subjects - Significant subcutaneous fat above the knee as determined by circumference of 50cm
4. Generally considered healthy according to medical history, physical examination, ECG and laboratory evaluation with a special emphasis on metabolic parameters (fasting glucose concentration < 100 mg, normal blood pressure).
5. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
6. Subjects must sign an informed consent indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

1. Unable to tolerate subcutaneous injection.
2. Subjects with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders, that in the opinion of the investigator, put the subject at significant risk, are not eligible.
3. Positive blood screen for Hepatitis B surface antigen (HbSAg), Hepatitis C virus (HCV), or Human immunodeficiency virus (HIV), or positive urine screen for alcohol or drugs of abuse (unless prescribed by a physician).
4. Subjects with a clinical history of primary or secondary immunodeficiency, autoimmune disease or subjects taking immunosuppressive drugs such as corticosteroids are ineligible.
5. As a result of medical review, physical examination, the PI (or medically qualified nominee) considers the subject unfit for the study.
6. Known sensitivity to components of the injection formulation.
7. Prior wound, tattoo or infection in the treated area.
8. Prior invasive treatment such as surgery or injectable drug at the RZL-012 injected area.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — For lipedema - women only. For lipedema and Dercum- Post-menopausal women
Enrollment: 12 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 - Lipedema 60mg: Total dose of RZL-012 (mg) 60 Number of injections: 12
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
- Cohort 2 Lipedema 80mg: Total dose of RZL-012 (mg) 80 Number of injections: 16
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
Period: Overall Study
Arm/Group | Cohort 1 - Dercum's Disease | Cohort 2 - Lipedema 60mg | Cohort 2 Lipedema 80mg
Started | 6 | 3 | 3
Completed | 6 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2 - Lipedema 80mg: Total dose of RZL-012 (mg) 80 Number of injections: 16
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Dercum's Disease | Cohort 2 - Lipedema 60mg | Cohort 2 - Lipedema 80mg | Total
Number analyzed (Participants) | 6 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (6.3) | 57.3 (5.0) | 57.3 (5.0) | 57.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 5 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Any Grade 3 or Greater Event Intolerable Side Effect Experienced in a Cohort
Description: Trial will proceed as long as no more than one subject experiences an intolerable side effect in a cohort
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 Lipedema 80mg: Total dose of RZL-012 (mg) 80 Dose per Number of injections: 16
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
Arm/Group | Cohort 1 - Dercum's Disease | Cohort 2 - Lipedema 60mg | Cohort 2 Lipedema 80mg
Number analyzed (Participants) | 6 | 3 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 days
Groups:
- Cohort 2 - Lipedema 60 mg: Total dose of RZL-012 (mg) 60 Number of injections: 12,
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
- Cohort 2 - Lipedema 80 mg: Total dose of RZL-012 (mg) 80 Number of injections: 16
  RZL-012: The dosing regimen will be a single dose treatment injection of RZL-012 in multiple sites
Arm/Group | Cohort 1 - Dercum's Disease | Cohort 2 - Lipedema 60 mg | Cohort 2 - Lipedema 80 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Dercum's Disease (N=6) | Cohort 2 - Lipedema 60 mg (N=3) | Cohort 2 - Lipedema 80 mg (N=3)
Injection site pain (General disorders) | 2 | 2 | 1
pain (General disorders) | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03492840/Prot_002.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03492840/SAP_003.pdf